CLINICAL TRIAL: NCT00221741
Title: PLASMACARD - Fresh Frozen Plasma in Cardiac Surgery: Descriptive and Prognostic Study
Brief Title: Fresh Frozen Plasma in Cardiac Surgery: Descriptive and Prognostic Study
Acronym: PLASMACARD
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: 9293-02; 2002-006
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Heart Surgery; Blood Loss, Surgical
Keywords: Heart surgery; Blood Loss, Surgical; Mortality; Blood Transfusion; Cohort Studies
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fresh Frozen Plasma (blood product)

SUMMARY:
Despite experts' recommendations, the consumption of Fresh frozen plasma (FFP) is very heterogeneous among French cardiac surgery centers. This probably reflects heterogeneous practices that are not characterized and whose outcomes on morbidity and mortality are not documented.

The principal objective of the study is to describe transfusional strategies of FFP in patients undergoing cardiac surgery. The other objectives are: to assess the conformity of FFP transfusion or lack of transfusion to current French authorities' recommendations, to describe the post-operative mortality and morbidity and to assess the prognostic role of FFP on mortality and morbidity. Prognostic analyses will take into account other prognostic factors of mortality and morbidity.

1500 patients undergoing cardiac surgery and presenting with a serious bleeding (or transfused with FFP without bleeding) will be included in the study.

DETAILED DESCRIPTION:
Background

Fresh frozen plasma (FFP) transfusions recommendations are essentially based on experts' opinions. However, disparity in consumption of FFP by cardiac surgery centers in France probably reflects heterogeneous practices that are not well characterized. Furthermore, health outcomes of these strategies on morbidity and mortality are not documented.

Objectives

Primary: to describe transfusional strategies of FFP in patients undergoing cardiac surgery and either presenting a serious bleeding during pre, per or post-operative periods or transfused by FFP without a serious bleeding.

Secondary:

* To estimate the conformity of transfusion or lack of transfusion of FFP to French authorities recommendations.
* To describe the post-operative mortality and morbidity.
* To evaluate the prognostic role of FFP transfusion on mortality and morbidity

Study design

Prospective prognostic cohort study, with an exhaustive recruitment in participating cardiac surgery centers during the study period.

Eligibility criteria

Centers: 16 French cardiac surgery centers.

Patients:

* Coronary artery bypass grafting (CABG), valvular replacement, surgery for thoracic aorta aneurysm or dissection, heart graft.
* Serious bleeding or FFP transfusion during pre, per or post-operative period.
* Patient's consent for collecting medical data

Analysis

Descriptive analysis of transfusional strategies according to patients' characteristics, type of surgery and circumstances of transfusions.

Conformity to French authorities' current recommendations. Multivariate analysis of the prognostic role of FFP transfusion on 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass grafting (CABG), valvular replacement, surgery for thoracic aorta aneurysm or dissection, heart graft.
* Serious bleeding or FFP transfusion during pre, per or post-operative periods.
* Patient's consent for collecting medical data

Exclusion Criteria:

* Congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1497 (Actual)
Dates: Start 2004-02; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Puntous, Dr, Principal Investigator — University Hospital, Bordeaux; Gérard Janvier, Professor, Study Director — University Hospital, Bordeaux; Paul Perez, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Département d'anesthésie-réanimation II (DAR II), Hôpital Haut-Lévêque, Av de Magellan, Pessac, France